CLINICAL TRIAL: NCT03184857
Title: Two Stage Sinus Lifting Using Nano Hydroxyapatite Particles [Nanostreams] Versus Deprotenized Bovine Bone [Tutogen] : Randomized Clinical Trial.
Brief Title: Open Maxillary Sinus Augmentation Using Different Types of Bone Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Nour-El deen, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cebc.cairouniversity - 1025
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Maxillary Sinus Augmentation
Keywords: maxillary sinus; augmentation; bovine bone; Nano hydroxy appatite

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two stage sinus lifting using bovine bone particles (Active Comparator): Open maxillary sinus lifting will be done with sinus augmentation using bovine bone particles
  Interventions: Procedure: open maxillary sinus lifting
- two sage sinus lifting using Nano HA bone particles (Experimental): Open maxillary sinus lifting will be done with sinus augmentation using Nano HA bone particles
  Interventions: Procedure: open maxillary sinus lifting

INTERVENTIONS:
Procedure: open maxillary sinus lifting — biopsy of the region 6 months later

SUMMARY:
Two stage sinus lifting using Nano hydroxyapatite particles [Nanostreams] versus Deprotenized bovine bone [Tutogen] : Randomized clinical trial.

comparing between Height of new bone formation, Bone area percent( Histomorphometric)

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* sinus pathology
* heavy smokers
* patients with systemic disease uncontrolled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
histomorphometric analysis | 6 months
  histomorphometric analysis to measure new bone percent formation and residual bone graft percent

SECONDARY OUTCOMES:
new height of bone gained | 6 months
  CBCT 6 months postoperative to measure the new height of bone

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Ahmed Nour Eldeen, Cairo, Egypt

REFERENCES:
- [Derived] Nour M, Shawky M, Abaas RA, Hakam M, Atef M. Two Stage Sinus Lifting Using Nanohydroxyapatite Particles Versus Deproteinized Bovine Bone: Randomized Clinical Trial. Clin Implant Dent Relat Res. 2025 Feb;27(1):e13410. doi: 10.1111/cid.13410. Epub 2024 Oct 31. PMID 39478644